CLINICAL TRIAL: NCT02184533
Title: A Phase I Study Evaluating the Efficacy and Safety of Sodium Selenite in Combination With Palliative Radiation Therapy in Patients With Metastatic Cancer
Brief Title: Sodium Selenite and Radiation Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-30587; NCI-2014-01361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PROS0047 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer; Multiple Myeloma; Plasmacytoma
MeSH Terms: conditions — Prostatic Neoplasms; Multiple Myeloma; Plasmacytoma | interventions — Sodium Selenite; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sodium selenite and radiation therapy) (Experimental): Patients receive sodium selenite PO 2 hours before daily radiation therapy treatments. Treatment continues for the duration of the course of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sodium selenite; Radiation: radiation therapy; Other: laboratory biomarker analysis; Other: pharmacological study; Other: questionnaire administration

INTERVENTIONS:
Drug: sodium selenite — Given PO
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
The purpose of this study is to determine the maximum-tolerated dose (MTD) of sodium selenite when administered in combination with radiation therapy to subjects with metastatic cancer based on safety and tolerability.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the maximum tolerated dose (MTD) of sodium selenite when given in combination with palliative radiation therapy
* To assess the safety and tolerability of the combination of sodium selenite and palliative radiation therapy in metastatic cancer

Secondary Objectives:

* To assess the pharmacokinetics of sodium selenite
* To evaluate the anti tumor activity of sodium selenite and palliative radiation therapy when given in combination

OUTLINE:

Patients receive sodium selenite orally (PO) 2 hours before daily radiation therapy treatments. Treatment continues for the duration of the course of radiation therapy in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed adenocarcinoma of the prostate from a prostate biopsy or prostatectomy specimen (primary site), or histological confirmation of adenocarcinoma /carcinoma in a metastatic site of disease in the setting of elevated PSA and imaging consistent with metastatic prostate cancer, or history of prostate cancer with documented metastasis, or histologically confirmed other solid tumor malignancy, multiple myeloma, or plasmacytoma with pathological confirmation of metastasis
2. Metastatic cancer requiring palliative radiation therapy
3. For patients with metastatic prostate cancer, PSA ≥ 2 ng/mL, except for patients who have recently started androgen deprivation therapy with PSA < 2 ng/mL
4. Age ≥18 years
5. Life expectancy greater than 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 or Karnofsky performance status ≥ 80%
7. QT interval corrected using Fridericia's method (QTcF) < 460 msec (see Appendix C for Fredericia's criteria).
8. Ability to understand and the willingness to sign a written informed consent document

Exclusion criteria:

1. Inadequate organ function, as evidenced by any of the following at screening:

   * Absolute neutrophil count (ANC) < 1500/µL
   * Platelet count ≤ 100 x 109/L
   * Serum creatinine > 2.0 mg/dL
   * Total bilirubin > 1.5 x upper limit of normal (ULN)
   * AST, and/or ALT > 2 x ULN
   * Hemoglobin < 9 g/dL
2. Men with reproductive potential who do not agree to use an accepted and effective method of contraception during the study treatment period and for at least 3 months after completion of the study treatment
3. History of other malignancies within 5 years prior to Day 1 except for tumors that in the opinion of the investigators have a negligible risk for metastasis or death, such as (but not exclusively) adequately controlled basal cell carcinoma, squamous cell carcinoma of the skin, or early stage bladder cancer
4. Current, or recent (within 4 weeks of the first treatment of this study) cytotoxic chemotherapy (eg, cisplatin, taxol) or experimental drug therapy, or planned participation in an experimental drug study
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant vascular disease (eg, aortic aneurysm, aortic dissection), symptomatic peripheral vascular disease, or psychiatric illness/social situations that would limit compliance with study requirements
6. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
7. History of stroke or transient ischemic attack within 6 months prior to study enrollment
8. The subject is known to be positive for the human immunodeficiency virus (HIV) and is receiving antiretroviral therapies. Subjects known to be HIV positive who do not require antiretroviral therapy will be eligible if they meet other entry criteria
9. Women who are pregnant or breastfeeding
10. Inability to comply with study and/or follow up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
MTD defined as the maximum dose at which =< 1 of 3 to 6 subjects in a dose group experience a drug-related dose-limiting toxicity, graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version (v)4.0 | 3 weeks
Safety and tolerability of the combination using the NCI Common Toxicity Criteria v4.0 grading system for adverse events | Up to 2 years
  Safety observations and measurements including adverse events, laboratory data, vital signs, and performance status will be summarized.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile | Week 1, day 1: at predose; 15 minutes; and at 1, 2, 4, and 24 hours; weeks 2 and 4, day 1: at predose and 1 hour
  PK parameters will be calculated using non-compartmental and/or compartmental models and PK parameters (if possible, maximum concentration [Cmax], time to Cmax, area under the curve during the dosing interval, half-life, oral clearance) will be summarized and presented.
Overall biochemical response rate | Up to 11 weeks
  Biochemical response defined as PSA decline >= 50% from baseline at 8 weeks of therapy and which has been confirmed with a second PSA at >= 3 weeks later.
Tumor responses within the radiation therapy field, assessed using Response Evaluation Criteria in Solid Tumors 1.1 | Up to 2 years
Response rate (complete response, partial response and stable disease) within the radiation therapy field | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Knox, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No